CLINICAL TRIAL: NCT05645198
Title: The Effect of Carboxymetyl Starch (Oozfix) on Preventing Postoperative Complication After Gastrectomy: Single-center, Non-inferiority, Open-label Randomized Trial
Brief Title: The Effect of Carboxymetyl Starch (Oozfix) on Preventing Postoperative Complication After Gastrectomy
Acronym: OOZFIX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bucheon St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Hayemin Lee, Assistant Professor, Bucheon St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HC22DISC0039
Record Dates: First submitted 2022-11-15; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — Diagnosis-Related Groups; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oozfix (Experimental): Arm with oozfix after gastrectomy
  Interventions: Drug: Oozfix
- Greenplast (Active Comparator): Arm with greenplast after gastrectomy
  Interventions: Drug: Greenplast

INTERVENTIONS:
Drug: Oozfix — Directly apply carboxymetyl starch (Oozfix) 5 gram evenly at the suprapancreatic surgical bed after gastrectomy
  Other Names: Case group
  Arms: Oozfix
Drug: Greenplast — Directly apply Greenplast (Aprotinin 1000kIU/mL, Thrombin 500IU/mL, Fibrinogen 95mg/mL) 4 gram evenly at the suprapancreatic surgical bed after gastrectomy
  Other Names: Control Group
  Arms: Greenplast

SUMMARY:
Although the technique of radical gastrectomy had been advanced, postoperative complication can occur in 13~25% of patient after radical gastrectomy. Pancreatic fistula and postoperative bleeding was reported as 2~30% and 1~2%, respectively. These complications often result fatal clinical course, so localized fibrin agent has been widely used at postoperative surgical bed after radical gastrectomy.

Recently, natural origin polysaccharide-based carboxymetyl starch was approved as localized coagulative, no well-designed report was adressed in gastric cancer surgery field. This agent can formate physical barrier after application, thus can prevent microbleeding or pancreatic fistula after gastrectomy. THIS study is single-center, non-inferiority, open-label randomized trial that evaluates the effect of carboxymetyl starch (Oozfix) on preventing postoperative complication after gastrectomy.

DETAILED DESCRIPTION:
Although the technique of radical gastrectomy had been advanced, postoperative complication can occur in 13~25% of patient after radical gastrectomy. Pancreatic fistula and postoperative bleeding was reported as 2~30% and 1~2%, respectively. These complications often result fatal clinical course, so localized fibrin agent has been widely used at postoperative surgical bed after radical gastrectomy.

Recently, natural origin polysaccharide-based carboxymetyl starch was approved as localized coagulative, no well-designed report was adressed in gastric cancer surgery field. This agent can formate physical barrier after application, thus can prevent microbleeding or pancreatic fistula after gastrectomy. THIS study is single-center, non-inferiority, open-label randomized trial that evaluates the effect of carboxymetyl starch (Oozfix) on preventing postoperative complication after gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Gastric adenocarcinoma patient who underwent radical gastrectomy at Bucheon St. Mary's Hospital
2. Patient's Age is above 19 and less than 80
3. ECOG performance score : 0~2

Exclusion Criteria:

1. Patient who underwent emergent gastrectomy
2. Patient who requires palliative gastrectomy due to advanced or metastatic carcinoma
3. Patient who requires operation due to other malignancy other than adenocrcinoma
4. Patient who underwent emergent gastrectomy or pancreatectomy before this study
5. Patient who underwent chemoradiation
6. Patient who took anticoagulants or with coagulopathy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of (patient who suffers from) pancreatic fistula | Postoperative day 3
  Ratio of patient who suffers from pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Hayemin LEE, Study Chair — Bucheon St. Mary's Hospital
Locations (1):
- BucheonStMarys, Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Washio M, Yamashita K, Niihara M, Hosoda K, Hiki N. Postoperative pancreatic fistula after gastrectomy for gastric cancer. Ann Gastroenterol Surg. 2020 Sep 21;4(6):618-627. doi: 10.1002/ags3.12398. eCollection 2020 Nov. PMID 33319151